CLINICAL TRIAL: NCT04782999
Title: Effect of RYGB on Alpha- and Beta Cell Function and Sensitivity to Incretins in Patients With Type 2 Diabetes
Acronym: BETASIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Maria Saur Svane, MD, PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: H-7-2014-010
Record Dates: First submitted 2021-02-26; First posted 2021-03-04 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Type2 Diabetes; Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Glucose Tolerance Test

STUDY DESIGN:
Intervention Model Description: Prospective evaluation of gastric bypass patients, who will be examined before, 1 week and 3 months after the gastric bypass operation.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oral glucose tolerance test (Active Comparator): Oral glucose tolerance test with ingestion of 75 g glucose and blood sampling.
  This test will be performed before and 3 months after RYGB.
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test
- Hyperglycemic clamp with saline infusion combined with arginine test (Active Comparator): Hyperglycemic clamp with blood glucose kept at 15 mmol/L by adjustable infusions of intraveneous glucose for 120 min with co-infusion of saline.
  After 120 min an arginine test with infusion of 50 g Arginine is performed.
  This test will be performed before, 1 week and 3 months after RYGB.
  Interventions: Diagnostic Test: Hyperglycemic clamp with infusion of saline, GLP-1 or GIP
- Hyperglycemic clamp with GLP-1 infusion (Active Comparator): Hyperglycemic clamp with blood glucose kept at 15 mmol/L by adjustable infusion of intraveneous glucose for 90 min with co-infusion of GLP-1.
  This test will be performed before, 1 week and 3 months after RYGB.
  Interventions: Diagnostic Test: Hyperglycemic clamp with infusion of saline, GLP-1 or GIP
- Hyperglycemic clamp with GIP infusion (Active Comparator): Hyperglycemic clamp with blood glucose kept at 15 mmol/L by adjustable infusions of intraveneous glucose for 90 minutes with co-infusion of GIP.
  This test will be performed before, 1 week and 3 months after RYGB.
  Interventions: Diagnostic Test: Hyperglycemic clamp with infusion of saline, GLP-1 or GIP

INTERVENTIONS:
Diagnostic Test: Oral Glucose Tolerance Test — Standard test of glucose tolerance with ingestion of 75 g glucose followed by blood sampling.
  Arms: Oral glucose tolerance test
Diagnostic Test: Hyperglycemic clamp with infusion of saline, GLP-1 or GIP — Blood glucose kept at 15 mmol/L via iv 20% glucose infusions.
  Primed co-infusion of either:
  * Saline
  * GLP-1 (Prime dose 6 pmol/kg, infusion 1 pmol/kg/min)
  * GIP (Prime dose 3 pmol/kg, infusion 1.5 pmol/kg/min).
  Arms: Hyperglycemic clamp with GIP infusion; Hyperglycemic clamp with GLP-1 infusion; Hyperglycemic clamp with saline infusion combined with arginine test

SUMMARY:
The aim of the study is to investigate the effect of Roux-en-Y gastric bypass (RYGB) on pancreatic alpha and beta-cell function and for the sensitivity of incretin hormones in patients with pre-operative type 2 diabetes.

Primary hypotheses:

* After RYGB, the sensitivity to GLP-1 and GIP is improved (improved insulinotropic effect).
* After RYGB, the insulin secretion improves during an oral glucose tolerance test within 3 months postoperatively.
* After RYGB, the insulin secretion during intraveneous stimulation with glucose or non-glucose (arginin) is unchanged.

DETAILED DESCRIPTION:
Design: 12 patients with type 2 diabetes will be recruited.

All subjects will undergo 11 study visits: four visits before, three visits at 1 week after surgery and four visits at 3 months postoperatively:

* Oral glucose tolerance tests (OGTTs) with measurement of GLP-1 and GIP secretion will be performed before and 3 months post-surgery.
* Hyperglycemic clamps with co-infusion of saline, GLP-1 or GIP will be performed in a randomised order at three separate study visits in randomized order before, 1 week and 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for RYGB in Denmark (ie. BMI > 35 in the presence of obesity related co-morbidities as type 2 diabetes)
* Type 2 diabetes
* Pre-operative: Fasting plasma glucose ≥7,0 mmol/L or 2 hour plasma glucose ≥ 11,1 mmol/L (after pausing antidiabetic medication for a minimum of 3 days)
* Written informed consent.

Exclusion Criteria:

* Exclusion criteria for RYGB (psychiatric illness, obesity triggered by medical treatment for psychiatric illness, mental retardation, alcohol or drug abuse, severe heart-lung disease despite optimal medical treatment, previous serious problems with universal anesthesia, previous peritonitis, large hiatus hernia, diseases of the ventricle / previously complicated upper abdominal surgery, recurrent esophagitis, poor compliance).
* Type 2 diabetes where antidiabetic medication cannot be paused for 3 days.
* Pregnancy and breast-feeding.
* Hemoglobin <7.0 mmol/L

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Insulinotropic effects of GLP-1 and GIP | Change from before to 1 week and 3 months after RYGB
  Insulin secretion during steady state of all hyperglycemic clamps
Insulin secretion during oral stimulation | Change from before to 3 month after RYGB
  AUC of C-peptide during oral glucose tolerance test
Insulin secretion during iv stimulation | Change from before to 1 week and 3 months after RYGB
  Insulin secretion during hyperglycemic clamp with saline infusion and during argininine iv stimulation test

SECONDARY OUTCOMES:
Alpha cell function | Change from before to after 1 week and 3 months after RYGB
  Glucagon secretion during hyperglycemic clamps

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No